CLINICAL TRIAL: NCT07045896
Title: Fucoidan Therapy in Adults With Active Rheumatoid Arthritis and Inadequate Response to Conventional DMARDs: a Single Center, Randomised, Double-blind, Placebo-controlled, Phase 2 Trial
Brief Title: Fucoidan in the Treatment of Active Rheumatoid Arthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Fanlei Hu, Professor, Department of Rheumatology and Immunology, Peking University People's Hospital, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024PHB505-001
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-01

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — fucoidan; Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fucoidan Add-on Therapy (Experimental): On the basis of the original conventional treatment regimen, 2000 mg of fucoidan was administered orally twice a day for 12 weeks.
  Interventions: Drug: Fucoidan
- Placebo Add-on Therapy (Placebo Comparator): On the basis of the original conventional treatment regimen, 2000 mg of placebo was administered orally twice a day for 12 weeks.
  Interventions: Drug: Corn starch

INTERVENTIONS:
Drug: Fucoidan — Background Therapy: Continued pre-existing conventional RA treatment at stable doses Intervention: Oral fucoidan Dosage Form: Size-0 gelatin capsules containing 1000mg fucoidan powder Dosage: 2000mg (2 capsules) per dose, twice daily (BID) Duration: 12 weeks continuous treatment
  Arms: Fucoidan Add-on Therapy
Drug: Corn starch — Background Therapy: Continued pre-existing conventional RA treatment at stable doses Intervention: Oral Corn starch as Placebo Dosage Form: Size-0 gelatin capsules containing 1000mg Placebo powder Dosage: 2000mg (2 capsules) per dose, twice daily (BID) Duration: 12 weeks continuous treatment
  Arms: Placebo Add-on Therapy

SUMMARY:
Rheumatoid arthritis (RA) is a chronic autoimmune disease characterized by joint destruction and autoantibody production. Scavenger receptor-A (SR-A), a pattern recognition receptor primarily expressed on myeloid-derived cells, is significantly elevated in the serum of RA patients. Genetic knockout of SR-A completely protects mice from collagen-induced arthritis (CIA). As an SR-A inhibitor, fucoidan markedly suppresses the progression of CIA in mice. Given the potential role of SR-A in RA pathogenesis, the investigators hypothesize that fucoidan may exert therapeutic effects in RA by specifically targeting human SR-A.

This study aims to investigate the efficacy of fucoidan in RA treatment through a randomized, double-blind, placebo-controlled trial, providing original insights into its clinical application. The investigators plan to enroll 38 patients each in the fucoidan treatment group and the control group, with a 12-week follow-up period. Clinical manifestations, laboratory parameters, and disease activity will be systematically evaluated to assess therapeutic outcomes. The findings will provide evidence-based medical data for RA treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years (inclusive) at screening, regardless of gender, with a minimum weight of 35 kg.
* Patients meeting the 2010 ACR classification criteria for rheumatoid arthritis.
* Patients with active rheumatoid arthritis showing moderate-to-high disease activity (DAS28-ESR >3.2) despite current treatment.
* If receiving conventional NSAIDs or other pain medications, the dose must have been stable for at least 2 weeks prior to the first study drug administration and remain unchanged during the study period.
* If taking oral corticosteroids, patients must have been on treatment for at least 4 weeks, with the dose stabilized at an average of ≤1.0 mg/kg/day prednisone equivalent for at least 4 weeks prior to the first study drug administration, and remain unchanged during the study period.
* If receiving DMARDs (methotrexate ≤25 mg/week with folic acid supplementation [recommended ≥5 mg/week] or leflunomide ≤40 mg/day), patients must have been on treatment for ≥8 weeks, with the dose stable for at least 4 weeks prior to the first study drug administration, and remain unchanged during the study period.
* Female patients of childbearing potential must have negative serum and urine pregnancy test results at screening.
* From the time of signing the informed consent form throughout the study and for 3 months after the last dose, female patients of childbearing potential and male patients who have not undergone vasectomy must use effective contraception.
* Patients must be willing and able to comply with the study restrictions.
* Patients must sign the informed consent form, understand the purpose and procedures of the study, and be willing to participate in the study.

Exclusion Criteria:

* Patients currently receiving biologic therapy.
* Patients with other inflammatory joint diseases or connective tissue diseases.
* Patients with significant bone marrow impairment or significant anemia, leukopenia, or thrombocytopenia secondary to inactive rheumatoid arthritis.
* Patients with persistent or severe infections within 3 months prior to enrollment.
* Patients with uncontrolled hypertension, uncontrolled diabetes, unstable ischemic heart disease, active inflammatory bowel disease, active peptic ulcers, terminal illnesses, or other conditions that, in the investigator's opinion, would pose a risk to the patient's participation in the study.
* Patients with clinically relevant cardiovascular, hepatic, neurological, endocrine, or other major systemic diseases that would complicate the implementation of the protocol or interpretation of study results.
* Patients with severe hypoalbuminemia (serum albumin <30 g/L), such as due to severe liver disease or nephrotic syndrome.
* Patients with moderate or severe renal impairment, defined as serum creatinine >133 μmol/L (or 1.5 mg/dL).
* Patients with a recent or clinically significant history of drug or alcohol abuse.
* Patients with impaired liver function or persistent alanine aminotransferase levels >2 times the upper limit of normal.
* Pregnant patients.
* Breastfeeding patients.
* Patients with congenital or acquired severe immunodeficiency, a history of cancer or lymphoproliferative disorders, or those who have undergone total lymphoid irradiation.
* Patients with known HIV-positive status.
* Patients with known positive serology for hepatitis B or hepatitis C.
* Patients enrolled in any other clinical trial involving off-label use of investigational drugs or devices, or enrolled in any other type of medical research.
* Patients with any active infection (including chronic or localized infections) requiring antimicrobial therapy within 28 days prior to the first study drug dose.
* Patients with a body mass index (BMI) <18.5 kg/m² or >30 kg/m².

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients achieving the American College of Rheumatology 20% improvement criteria (ACR20) at Week 12. | at Week 12
  The ACR20 criteria for evaluating the condition are: a 20% or greater improvement in the number of tender joints compared to baseline, a 20% or greater improvement in the number of swollen joints, and a 20% or greater improvement in three of the following five core indicators: A) the patient's overall assessment of disease activity, B) the physician's overall assessment of disease activity, C) the patient's assessment of arthritis pain, D) Health Assessment Questionnaire Disability Index (HAQ-DI), and E) C-reactive protein (CRP) for assessing physical function.

SECONDARY OUTCOMES:
Proportion of patients achieving Disease Activity Score in 28 joints using Erythrocyte Sedimentation Rate (DAS28-ESR) remission or low disease activity at Week 12 | at Week 12
  DAS28-ESR remission: DAS28 <2.6; DAS28-ESR low disease activity: DAS28 ≤3.2
Change from baseline in Clinical Disease Activity Index (CDAI) and Simplified Disease Activity Index (SDAI) at Week 12 | at Week 12
  CDAI and SDAI indices assess rheumatoid arthritis disease activity through tender/swollen 28-joint counts, patient and physician global assessments (0-10 cm VAS), with SDAI additionally incorporating C-reactive protein (CRP) levels.
Percentage of patients achieving good or moderate EULAR response at Week 12 | at Week 12
  A good response is defined as DAS28-ESR ≤ 3.2, with a decrease of more than 1.2 from baseline; a moderate response is defined as meeting one of the following criteria: DAS28-ESR ≤ 3.2, with a decrease of more than 0.6 and no more than 1.2 from baseline; 3.2 <DAS28-ESR ≤ 5.1, with a decrease of more than 0.6 from baseline; DAS28-ESR> 5.1, with a decrease of more than 1.2 from baseline.
Proportion of subjects achieving American College of Rheumatology 50% improvement criteria (ACR50) at Week 12 | at Week 12
  The evaluation is based on: a 50% to 70% or greater improvement in the number of tender joints compared to baseline; a 50% to 70% or greater improvement in the number of swollen joints; and a 50% to 70% or greater improvement in three of the remaining five core indicators: the patient's overall assessment of disease activity, the physician's overall assessment of disease activity, the patient's assessment of arthritis pain, and the Health Assessment Questionnaire Disability Index (HAQ-DI) and C-reactive protein (CRP) for assessing physical function.
Percentage of participants meeting the 2011 ACR/EULAR Boolean remission criteria at Week 12 | at Week 12
  he simplified definition of ACR/EULAR remission criteria in 2011 was: Tender Joint Count <1; Swollen Joint Coun <1; overall disease activity assessment in ACR/EULAR patients <1; CRP <1mg/L

CONTACTS AND LOCATIONS:
Overall Officials: Fanlei Hu, Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li ZG. A new look at rheumatology in China--opportunities and challenges. Nat Rev Rheumatol. 2015 May;11(5):313-7. doi: 10.1038/nrrheum.2014.218. Epub 2015 Jan 20. PMID 25599919
- [Background] Hu F, Jiang X, Guo C, Li Y, Chen S, Zhang W, Du Y, Wang P, Zheng X, Fang X, Li X, Song J, Xie Y, Huang F, Xue J, Bai M, Jia Y, Liu X, Ren L, Zhang X, Guo J, Pan H, Su Y, Yi H, Ye H, Zuo D, Li J, Wu H, Wang Y, Li R, Liu L, Wang XY, Li Z. Scavenger receptor-A is a biomarker and effector of rheumatoid arthritis: A large-scale multicenter study. Nat Commun. 2020 Apr 20;11(1):1911. doi: 10.1038/s41467-020-15700-3. PMID 32312978
- [Background] Yeh CW, Shih CJ, Liu TC, Chiou YL. Effects of oligo-fucoidan on the immune response, inflammatory status and pulmonary function in patients with asthma: a randomized, double-blind, placebo-controlled trial. Sci Rep. 2022 Oct 28;12(1):18150. doi: 10.1038/s41598-022-21527-3. PMID 36307493
- [Background] Konic Ristic A, Ryan S, Attjioui M, O'Connell S, Gibney ER. Effects of an Extract of the Brown Seaweed Ascophylum nodosum on Postprandial Glycaemic Control in Healthy Subjects: A Randomized Controlled Study. Mar Drugs. 2023 May 31;21(6):337. doi: 10.3390/md21060337. PMID 37367662